CLINICAL TRIAL: NCT03308331
Title: HIV-1 and Brain Interaction on Smoking Comorbidity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We originally had a collaboration with a PI but he has left the University.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, L. Elliot Hong, MD, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00075780
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: HIV; nicotine; brain; smoking
MeSH Terms: conditions — Smoking | interventions — Smoking Devices; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- HIV-1 smokers (Experimental)
  Interventions: Other: Tobacco smoking and nicotine patch
- HIV-1 nonsmokers (No Intervention)
- Healthy control smokers (Active Comparator)
  Interventions: Other: Tobacco smoking and nicotine patch
- Healthy control nonsmokers (No Intervention)
- HIV-1 nonsmokers using nicotine patch (Active Comparator)
  Interventions: Other: Tobacco smoking and nicotine patch
- HIV-1 nonsmokers using placebo patch (No Intervention)
- Healthy control nonsmokers using nicotine patch (Active Comparator)
  Interventions: Other: Tobacco smoking and nicotine patch
- Healthy control nonsmokers using placebo patch (No Intervention)

INTERVENTIONS:
Other: Tobacco smoking and nicotine patch — Tobacco smoking at each participant's regular cigarette. Over-the-counter nicotine patch use
  Arms: HIV-1 nonsmokers using nicotine patch; HIV-1 smokers; Healthy control nonsmokers using nicotine patch; Healthy control smokers

SUMMARY:
People living with HIV-1 have high rates of cigarette smoking, which may be related to nicotinic interaction with HIV-1 infection and brain function levels. The proposed project aims to understand these pathways using translational brain imaging and HIV-1 reactivation studies. The study proposes a targeted nicotine-brain investigation of the nicotinic effects in HIV-1 infection from cellular to brain circuitry levels.

DETAILED DESCRIPTION:
Smoking remains the leading cause of preventable morbidity and mortality in the United States. The alarmingly high smoking rates and unsatisfactory performance of standard smoking cessation efforts in people living with HIV/AIDS (PLWH) interfere with the overall progress in the treatment of HIV-1 infection. Our understanding of nicotine addiction mechanisms in PLWH, and how they are related to and interact with HIV-1 neuropathology, is limited and thus hindering the development of more effective, targeted treatments. The study will directly address neurological complication of this HIV-associated comorbidity at the brain circuitry level using state-of-the-art imaging tools and methods.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between ages 18-60 in good health
2. Ability to give written informed consent
3. For people living with HIV: should be diagnosed with HIV two years or more and on ART two years or more
4. For people living with HIV: should have achieved virologic suppression (defined as viral loads of ≤ 200 copies/ml), and without current signs of reactivation

Exclusion Criteria:

1. Inability to sign informed consent
2. Unable to undergo MRI scanning due to metallic devices or objects (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or claustrophobic to the scanner
3. Any major medical illnesses to include, but not limited to, uncontrolled high blood pressure or high blood sugar, cardiovascular disease, asthma, peripheral vascular diseases, coagulopathies, history of superficial or deep vein thrombosis as per medical history
4. Current substance-induced psychiatric disorders
5. Significant alcohol or other drug use, other than nicotine dependence or marijuana use
6. Gross structural abnormalities and/or have a history of syncope
7. Positive urine pregnancy tests
8. Any neurological illnesses to include, but not limited to, seizure disorders, multiple sclerosis, movement disorders, or history of head trauma, CVA, CNS tumor,
9. For people living with HIV: having AIDS or non-AIDS-defining cancer or active CNS and other opportunistic disease
10. For people living with HIV: on active treatment of hepatitis C virus (HCV)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Functional and structural connectivity using magnetic resonance imaging (MRI) | one day
  Resting functional MRI and diffusion imaging MRI

SECONDARY OUTCOMES:
HIV-1 reactivation | one day
  HIV-1 viral protein p24 expression

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States